CLINICAL TRIAL: NCT00349830
Title: Development of Novel Serum Markers for Monitoring Response to Anti-Cancer Therapy
Brief Title: Novel Serum Markers for Monitoring Response to Anti-Cancer Therapy
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-13535; 77923 (Other: Stanford University Alternate IRB Approval Number); IRB-13535 (Other: Stanford IRB); VAR0006 (Other: OnCore); 5R01CA18829804 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Carcinomas (Including Squamous Cell and Adenocarcinoma); Neoplasms
MeSH Terms: conditions — Carcinoma; Adenocarcinoma; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood draw

SUMMARY:
The purpose of this study is to measure the levels of serum proteins and other biomarkers in cancer patients and in patients suspected of having cancer. We believe that some of these markers may be useful for confirming the diagnosis or for selecting patients for specific types of cancer therapies. These markers may also help to predict response to therapy, relapse after therapy, and survival after therapy.

DETAILED DESCRIPTION:
This is a blood serum collection study at Stanford University for patients with cancer at a variety of disease sites. The purpose of this study is to collect and store blood serum from patients before, during, and after anti-cancer therapy to find new biomarkers that signal disease or response to anti-cancer therapy. The collection and analysis of these biomarkers may lead to improved diagnostic and treatment therapies for certain cancers in the future. We are also interested in collecting blood serum from healthy individuals such as the spouses, relatives, and friends of cancer patients to obtain healthy controls for comparison

ELIGIBILITY:
1. Age > or = 18; for the samples collected under the NIH grant, no subjects below the age of 20 will be enrolled.
2. Prior diagnosis of cancer or suspected of having cancer
3. Karnofsky performance status of greater than 70
4. Standard pretreatment evaluation
5. Signed Stanford University Human Subjects Committee consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2002-01; Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for disease | Day one

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Diehn, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States